CLINICAL TRIAL: NCT00008164
Title: Transplantation Using Umbilical Cord And Placental Blood
Brief Title: Umbilical Cord Blood and Placental Blood Transplantation in Treating Patients With Hematologic Cancer or Aplastic Anemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068384; CPMC-IRB-7934; CPMC-CAMP-021; NCI-G00-1899
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-01

CONDITIONS: Childhood Langerhans Cell Histiocytosis; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; childhood Langerhans cell histiocytosis; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; recurrent/refractory childhood Hodgkin lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Recurrence; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Cord Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Umbilical cord blood or placental blood transplantation may be able to replace immune cells that were destroyed by the chemotherapy or radiation therapy that was used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of umbilical cord blood and placental blood transplantation in treating patients who have hematologic cancer or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with chronic myeloid leukemia, acute leukemia, lymphoma, myeloma, myelodysplasia, aplastic anemia, Fanconi's anemia, histiocytosis, hereditary immunodeficiency, or storage disorder treated with allogeneic umbilical cord and placental blood transplantation.
* Determine the toxicity of this regimen in these patients.
* Determine survival in these patients treated with this regimen.
* Determine the incidence of graft-versus-host disease in these patients treated with this regimen.

OUTLINE: Patients receive a standard preparative regimen for their disease. Following the preparative regimen patients undergo umbilical cord blood stem cell transplantation on day 0.

Patients are followed every 1-2 weeks for 6 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myeloid leukemia, acute leukemia, lymphoma, myeloma, myelodysplasia, aplastic anemia, Fanconi's anemia, histiocytosis, hereditary immunodeficiency, or storage disorder
* Eligible for allogeneic bone marrow transplantation, but lacking a donor
* Available donor umbilical cord blood that is mismatched on no more than 2 HLA loci

  * HIV negative
  * Hepatitis B surface antigen and hepatitis C negative

PATIENT CHARACTERISTICS:

Age:

* Under physiologic 60

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 times normal
* No severe hepatic disease
* Hepatitis B surface antigen and hepatitis C negative

Renal:

* Creatinine less than 2 times normal

Other:

* HIV negative
* Not pregnant or nursing
* No other serious medical or psychiatric illness that would preclude study compliance
* No serious infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-01

PRIMARY OUTCOMES:
Response rate
Toxicity
Survival
Incidence of graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: David G. Savage, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States

REFERENCES:
- [Result] Styczynski J, Cheung YK, Garvin J, Savage DG, Billote GB, Harrison L, Skerrett D, Wolownik K, Wischhover C, Hawks R, Bradley MB, Del Toro G, George D, Yamashiro D, van de Ven C, Cairo MS. Outcomes of unrelated cord blood transplantation in pediatric recipients. Bone Marrow Transplant. 2004 Jul;34(2):129-36. doi: 10.1038/sj.bmt.1704537. PMID 15107815